CLINICAL TRIAL: NCT06650033
Title: Pelvis Adaptive Radiation Therapy
Brief Title: Pelvis Adaptive Radiotherapy (ART)
Acronym: Pelvis ART
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Royal North Shore Hospital (Other)
Collaborators: Northern Sydney and Central Coast Area Health Service (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pelvis Adaptive Radiotherapy
Record Dates: First submitted 2024-10-17; First posted 2024-10-21 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Pelvis Neoplasms
MeSH Terms: conditions — Pelvic Neoplasms | interventions — Radiotherapy, Image-Guided

STUDY DESIGN:
Intervention Model Description: Patients will be randomised to Adaptive radiotherapy or standard radiotherapy, 2:1 randomisation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adaptive radiotherapy +/- margin reduction (Active Comparator): Phase 1 and 2: Treating Radiation Therapists (RTs) on the treatment machine will review the treatment target and organs at risk contours that are automatically generated on the plan of the day. They will modify these safely, as required, and then also approve the computer generated re-plan of the day, within the bounds of departmental protocols and decision guides (RT led).
  Phase 2 only: Margin reduction facilitated by adaptive radiotherapy.
  Interventions: Radiation: Adaptive radiotherapy +/- margin reduction
- Standard radiotherapy (Active Comparator): Patients will receive standard image guided radiotherapy
  Interventions: Radiation: Image guided radiotherapy

INTERVENTIONS:
Radiation: Adaptive radiotherapy +/- margin reduction — Radiotherapy using adaptive technology to recontour and re-plan daily as required. Reductions in the PTV margin will also be introduced in the second phase of this study.
  Arms: Adaptive radiotherapy +/- margin reduction
Radiation: Image guided radiotherapy — Standard radiation treatment used in the department of radiation oncology for cancer in pelvic area
  Arms: Standard radiotherapy

SUMMARY:
Pelvis Adaptive radiotherapy (ART) is a two phase study looking at using adaptive radiotherapy to help reduce toxicity for cancer patients having radiotherapy in the pelvic region.

Adaptive radiotherapy is a new technology that provides the ability to account for daily changes in anatomy. Adaptive radiotherapy also provides a foundation for which radiotherapy margins might be safely reduced.

Phase 1 of this study is looking to see if a radiation therapist centred adaptive workflow can be implemented. If phase 1 of this study is safe and feasible, the study will proceed to phase 2. Phase 2 of the study looks at using adaptive technology to reduce radiation treatment margins. The primary aim of this study is to see whether margin reduced treatment using adaptive radiotherapy can reduce side effects for patients with cancer in the pelvic area.

DETAILED DESCRIPTION:
Despite major technological advancements in the delivery of pelvic radiation therapy including the use of dynamic therapy, image guidance, integrated boosting and stereotactic techniques, toxicity from pelvic radiation remains a significant issue impacting on patient's quality of life and preventing the delivery of higher (and more curative) doses of radiation. Although evidence showed that adaptive radiotherapy demonstrating promising reduction of acute toxicity, the uptake of adaptive radiotherapy remains poor as adaptive radiation therapy is very labour intensive, time consuming and usually requires a radiation oncologist (RO) and Medical Physicist in attendance to review/modify target contours. These practices of daily multi-disciplinary team (MDT) in person attendance is not sustainable in the long term. Since 2021, Royal North Shore Hospital has been treating patients with cancer in the pelvic with Adaptive Radiation Therapy (ART) and Radiation Therapists (RT) at the site have undergone a rigorous University based Advanced Practitioner training programme. This study aims to evaluate RT-led ART in a randomised trial to assess the safety and feasibility of ART in a two stage phase 3 randomised controlled trial.

If this study can prove safety and feasibility in the first phase, it will proceed to the second phase of the study which will look at using adaptive radiotherapy to safely reduce CTV and PTV margins. The primary aim of the study will be to measure the difference in combined acute patient reported gastrointestinal (GI) and genitourinary (GU) toxicity between ART with margin reduction versus standard radiotherapy. Secondary aims will be to look at differences in clinician and patient reported acute and late GI and GU toxicity, disease free survival locoregional control, location of recurrence, the efficiency of ART including time taken per treatment, radiation dosimetric differences between the treatment arms and patients' perception of ART.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18
2. ECOG performance status 0-2
3. Patients receiving curative or adjuvant pelvic radiation including:

   1. Prostate cancer where nodal treatment is required
   2. Prostate cancer post prostatectomy
   3. Bladder cancer
   4. Rectal cancer
   5. Anal cancer
   6. Adjuvant radiotherapy for gynaecological cancers
   7. Pelvic Lymph nodes only
4. Ability to understand and the willingness to sign an informed consent

Exclusion Criteria:

* Hip prosthesis
* Patient separation from approximate radiation centre to skin edge > 24cm, measured on diagnostic scan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2025-10-09 (Actual); Primary Completion 2029-11-30 (Estimated); Study Completion 2031-11-30 (Estimated)

PRIMARY OUTCOMES:
Dose coverage of Clinical Target Volume (CTV) (% of CTV receiving 95% of prescribed dose) will be performed between the two arms (Safety). | 12 months
  The CTV dose coverage must be equal or better in 90% of fractions for 90% of patients in the adaptive arm will be compared with the virtual image guided radiotherapy (IGRT) fraction. Dose coverage will be calculated as the percent of CTV receiving at least 95% of the prescribed dose (TD). Percentage will be measured from 0-100%, a higher % is a better outcome.
The percentage of organ at risk (OAR) dose volume histogram (DVH) metrics satisfying departmental protocol constraints will be compared for each patient between the two arms (Safety). | 12 months
  The OAR DVH dose constraints must be equal or better in 90% of fractions for 90% of patients compared with the virtual image guided radiotherapy (IGRT) fraction (safety). Percentage will be measured from 0-100%, a higher % is a better outcome.
The percentage of successfully delivered fractions on the adaptive arm will be measured (feasibility). | 12 months
  At least 90% of patients must have 90% of planned adaptive treatments successfully delivered in phase 1 of the study. Percentage will be measured from 0-100%, a higher % is a better outcome.
Acute patient reported toxicity | Within 90 days of patients completing treatment
  The study will measure the difference in patient reported combined maximum genitourinGU and GI toxicity (Grade 2 or higher) as per PRO-CTCAE between the two treatment arms. PRO-CTCAE scale is generally measured from 0 to 5, higher scale being a worse outcome.

SECONDARY OUTCOMES:
Acute clinician reported toxicity | Within 90 days of patients completing treatment
  The study will measure the difference in acute combined maximum genitourinary (GU) and gastroenterology (GI) toxicity (Grade 2 or higher) grading between the two treatment arms as reported by clinicians using CTCAE v5.0. The CTCAE scale is generally measured from 0 to 5, higher scale being a worse outcome.
Late clinician reported toxicity | 5 years
  The study will measure the difference in late GU and GI toxicity (Grade 2 or higher) between the two treatment arms as reported by clinicians using CTCAE v5.0. The CTCAE scale is generally measured from 0 to 5, higher scale being a worse outcome.
Late patient reported toxicity | 5 years
  The study will measure the difference in patient reported late GU and GI toxicity (Grade 2 or higher) between the two treatment arms as per PRO-CTCAE. The PRO-CTCAE scale is generally measured from 0 to 5, higher scale being a worse outcome.
Disease free survival (DFS) (incorporating biochemical DFS for prostate cancer patients | 5 years
  The rate of disease free survival and the rate of biochemical failure in prostate cancer as defined as Nadir+2.0, commencement of ADT for relapse or evidence of disease recurrence on imaging. DFS is measured as a continuous variable, a longer DFS is associated with better outcomes.
Time differences between treatment arms | 5 years
  The study will assess the average absolute treatment time difference per fraction for adaptive radiation therapy compared to standard IGRT. Time is measured as a continuous variable, this is a descriptive statistic and longer or shorter time is not necessarily better or worse.
Radiation dosimetric differences between treatment arms | 5 years
  The study will evaluate the radiation dosimetric differences between treatment using ART and treatment using standard IGRT.
Patient reported attitudes and perceptions | 1 and 5 years
  The study will assess the patient experience with radiotherapy on a five item questionnaire that uses a five-point Likert-scale (ranging from strongly disagree to strongly agree). Differences in responses for each question between the arms will be reported. Whether each perception is better or worse is dependent on the question.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Kneebone, Principal Investigator — Northern Sydney Local Health District
Locations (1):
- Northern Sydney Local Health District, St Leonards, New South Wales, Australia